CLINICAL TRIAL: NCT00058370
Title: A Trial Of Radioimmunotherapy, Reduced-Dose External Beam Craniospinal Radiation Therapy With IMRT Boost, And Chemotherapy For Patients With Standard-Risk Medulloblastoma
Brief Title: Intrathecal Radioimmunotherapy, Radiation Therapy, and Chemotherapy After Surgery in Treating Patients With Medulloblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-088; MSKCC-02088
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2019-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult medulloblastoma; untreated childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma | interventions — Cisplatin; Lomustine; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

ARMS (1):
- histologic proof of medulloblastoma (Experimental): This is a single-arm study of post-operative radioimmunotherapy (intrathecal 131-I-3F8), reduced-dose craniospinal radiation therapy (1800 cGy), primary site boost (to 5400 cGy) via IMRT and standard chemotherapy.
  Interventions: Drug: cisplatin; Drug: lomustine; Drug: vincristine sulfate; Procedure: adjuvant therapy; Radiation: iodine I 131 monoclonal antibody 3F8; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: lomustine
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: iodine I 131 monoclonal antibody 3F8
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radioimmunotherapy uses radiolabeled monoclonal antibodies to locate tumor cells and deliver radioactive tumor-killing substances to them without harming normal cells. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining intrathecal radioimmunotherapy and radiation therapy with combination chemotherapy may kill any tumor cells remaining after surgery.

PURPOSE: Phase II trial to study the effectiveness of combining intrathecal radioimmunotherapy and radiation therapy with combination chemotherapy in treating patients who have undergone surgery for medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of combining post-operative intrathecal radioimmunotherapy, craniospinal radiotherapy with intensity-modulated radiotherapy boost, and chemotherapy in patients with standard-risk medulloblastoma.
* Determine whether this regimen can maintain or exceed the current progression-free survival rate while decreasing long-term serious morbidity in these patients.
* Determine the long-term morbidities, most specifically neuropsychological, neuroendocrine, audiometric, and growth outcomes, in patients treated with this regimen.

OUTLINE:

* Radioimmunotherapy: Patients receive intrathecal iodine I 131 monoclonal antibody 3F8 on days 1 and 8.
* Radiotherapy: Beginning as soon as possible after radioimmunotherapy, patients undergo external-beam and intensity-modulated radiotherapy 5 days a week for 6 weeks.
* Chemotherapy: Patients receive vincristine IV once weekly for 8 weeks concurrently with radiotherapy. Beginning about 6 weeks after completion of radiotherapy (4 weeks after vincristine), patients receive cisplatin IV over 6 hours and oral lomustine on day 0 and vincristine IV on days 0, 7, and 14. Treatment repeats every 6 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 6-20 patients will be accrued for this study within 3.2 years.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must have histologic proof of medulloblastoma reviewed by the Department of Pathology at the Memorial Sloan-Kettering Cancer Center.
* Patients must begin study prescribed therapy within 42 days of neurosurgical resection of the tumor
* Age ≥ 3-years-old. Post-operative head MRI must confirm ≤ 1.5 cm2 of residual tumor is present.
* Head and spine MRI and lumbar CSF cytology must not show any definitive evidence of leptomeningeal dissemination (Chang stage M-0).
* Examinations evaluating extra-neural sites will not be mandated, but any performed for clinical indications must be free of metastatic disease.
* No prior RT or chemotherapy for the medulloblastoma is permitted Patients must have adequate CSF flow (defined as lack of compartmentalization) on an 111-Indium DTPA flow study.
* Patients must have adequate organ function as defined by:
* Hepatic: total bilirubin < 2.0 mg/dl, AST < 3 x the upper limit of normal.
* Renal: Calculated creatinine clearance or nuclear GFR ≥ 70 ml/min/1.73 m^2.
* The patient, or for minors, a parent or legal guardian, must give informed written consent indicating they are aware of the investigational nature of this study.

EXCLUSION CRITERIA:

* Unable to start study prescribed therapy within 42 days of neurosurgical resection of the tumor
* Age less than 3 years > 1.5 cm2 residual tumor on post-operative head MRI
* Evidence of leptomeningeal dissemination on head or spine MRI or CSF cytology positivity
* Evidence of extra-neural metastases
* Prior radiation therapy or chemotherapy for the medulloblastoma
* Inadequate CSF flow on 111-Indium DTPA flow study Patients with signs or symptoms suggestive of increased intracranial pressure (headache, emesis, ocular paresis) will not be eligible until they are cleared by neurology and/or neurosurgery.
* Pregnancy
* Total bilirubin ≥ 2.0 mg/dl
* AST ≥ 3 x the upper limit of normal
* Creatinine clearance and GFR < 70 ml/min/1.73 m^2

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Dunkel, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Histologic Proof of Medulloblastoma
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Histologic Proof of Medulloblastoma
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 6 [4 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility
Time Frame: 2 years
Population: No data were collected
Arm/Group | Histologic Proof of Medulloblastoma
Number analyzed (Participants) | 0

2. Primary Outcome: Progression-free Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Histologic Proof of Medulloblastoma
Number analyzed (Participants) | 0

3. Primary Outcome: Morbidity
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Histologic Proof of Medulloblastoma
Number analyzed (Participants) | 6
Participants
  Deceased | 3
  Alive | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Histologic Proof of Medulloblastoma
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Histologic Proof of Medulloblastoma (N=6)
Constipation (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Infection w.out neutropenia (Infections and infestations) | 2
Leukocytes (Investigations) | 1
Lymphopenia (Investigations) | 1
Neutrophils/gran (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Histologic Proof of Medulloblastoma (N=6)
Nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Fever (General disorders) | 2
Headache (Nervous system disorders) | 2
Pain, other (General disorders) | 2
Stomatitis/pharyn (Gastrointestinal disorders) | 2
Abdominal pain/cramping (Gastrointestinal disorders) | 1
Allergic Reaction/Hyper (Immune system disorders) | 1
Ataxia (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Derm, skin other (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Mood alteration-anxiety (Psychiatric disorders) | 1
Mucositis/Rad (Gastrointestinal disorders) | 1
Neuropathy-motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Ocular-Vision other (Eye disorders) | 1
Rash, desquamation (Skin and subcutaneous tissue disorders) | 1
SGOT (AST) (Investigations) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-02-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT00058370/Prot_SAP_000.pdf